CLINICAL TRIAL: NCT05189119
Title: Study of Pressure Support Under Non-invasive Ventilation in the Early Diagnosis of Left Ventricular Failure During Acute Exaverbation of Chronic Obstructive Pulmonary Disease
Brief Title: Use of PARniv for Early Diagnosis of LVF in AECOPD
Status: Completed | Type: Observational
Sponsor: University of Monastir (Other)
Responsible Party: Principal Investigator, Pr. Semir Nouira, professor, University of Monastir
Other Study IDs: pressure support /LVF/ AECOPD
Record Dates: First submitted 2021-12-27; First posted 2022-01-12 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Acute Heart Failure; COPD Exacerbation
Keywords: COPD; Left Ventricular Failure; Pressure Support under NIV
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- LVFgroup: patients with AECOPD and left ventricular failure
  Interventions: Diagnostic Test: non invasive ventilation
- non LVF group: patients with AECOPD and whithout left ventricular failure
  Interventions: Diagnostic Test: non invasive ventilation

INTERVENTIONS:
Diagnostic Test: non invasive ventilation — invasive mechanical ventilation session in the BIPAP Mode with a pressure support (PS) level of 5cmH2O, a positive end expiratory pressure (PEEP) level of 5 cmH2O and an inspiratory fraction of oxygen (FiO2) allowing a pulse saturation (SpO2) of at least 92% for a one minute and followed by an increase of the PS level to 30cmH2O.The plethysmographic PAR (PAR) was calculated based on the following formula: PARpleth= PP30 / PP5
  Other Names: NIV

SUMMARY:
Left ventricular failure (LVF) is a common cause of acute exacerbation of chronic obstructive pulmonary disease (AECOPD).

This association is frequently underestimated with regard to the difficulty of clinical diagnosis .

The investigators expect that the application of pressure support under NIV could be useful in this issue.

DETAILED DESCRIPTION:
Acute heart failure (AHF) is a common cause of COPD exacerbation however its role is very often underestimated. Until now, the use of echocardiography and some invasive hemodynamic exploration techniques such as the Swan-ganz catheter has been stated as reference. Other noninvasive diagnostic methods have been studied, such as systolic time intervals and Valsalva maneuver, but their application still difficult in patients with COPD exacerbation, especially in emergency department (ED) settings. the study aimed to evaluate the performance of a new diagnostic technique based on the measurement of the PAR using non invasive ventilation (NIV) for the early identification of left ventricular failure (LVF) in patients presenting to the ED with acute COPD exacerbation

ELIGIBILITY:
Inclusion Criteria:

* patients with a history of COPD
* consulted the emergency department for AECOPD defined by a respiratory rate >25c/min, SaO2 <90%, pH <7.35 and PaCO2 >6kPa were included.

Exclusion Criteria:

* hemodynamic instability requiring the use of vasoactive drugs
* patients with contraindications to NIV (Glasgow score <12, swallowing disorder or severe bronchial obstruction, vomiting, and those with upper airway obstruction or ongoing upper gastrointestinal bleeding and altered bronchial clearance)
* non cooperative patients
* who refused to give consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all patients presenting to the ED with an acute COPD exacerbation
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2022-01-03 (Actual); Primary Completion 2022-05-03 (Actual); Study Completion 2022-05-03 (Actual)

PRIMARY OUTCOMES:
left ventricular dysfunction | 24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- University hospital of Monastir, Monastir, Tunisia

REFERENCES:
- [Derived] Bel Haj Ali K, Sekma A, Chamtouri I, Beltaief K, Msolli MA, Mezgar Z, Bouida W, Boukef R, Boubaker H, Grissa MH, Nouira S. Pulse amplitude ratio under noninvasive ventilation as a new method in the diagnosis of left heart failure in patients with acute exacerbation of chronic obstructive pulmonary disease. BMC Cardiovasc Disord. 2023 Feb 24;23(1):105. doi: 10.1186/s12872-023-03089-y. PMID 36829108